CLINICAL TRIAL: NCT02350049
Title: Cementless Oxford Partial Knee Retrospective and Prospective Controlled Multi-center Observational Study
Brief Title: Cementless Oxford Partial Knee Controlled Observational Study
Acronym: GK10
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GK10
Record Dates: First submitted 2014-07-15; First posted 2015-01-29 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Investigational: Cementless Medial Partial Knee
- Control: Cemented Medial Partial Knee

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Cementless Oxford Partial Knee System.

DETAILED DESCRIPTION:
The study is designed to document and compare the clinical and radiographic results of the Cementless Oxford Partial Knee System (investigational device) to those of the cemented Oxford Partial Knee System (control device).

ELIGIBILITY:
Inclusion Criteria:

* have primary diagnosis of osteoarthritis or avascular necrosis limited to the medial compartment of the knee
* signed informed consent for patients contributing to investigational or control if required
* Male or female over the age of 21 years at the time of surgery
* Undergone primary partial knee arthroplasty as unilateral arthroplasty or bilateral arthroplasty, simultaneously or otherwise
* Patients that are current residents of the United Kingdom

Exclusion Criteria:

* Evidence of infection, sepsis, and osteomyelitis at the time of surgery
* Use in the lateral compartment of the knee
* Rheumatoid arthritis or other forms of inflammatory joint disease
* Revision of a failed prosthesis, failed upper tibial osteotomy or post-traumatic arthritis after tibial plateau fracture
* Insufficiency of the collateral, anterior, or posterior cruciate ligaments which would preclude stability of the device
* Partial or full thickness cartilage disease or damage to central part of the lateral femoral condyle
* Osteoporosis or insufficient bone stock
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infection which may spread to the implant site
* Rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram
* Vascular insufficiency, muscular atrophy, neuromuscular disease
* Incomplete or deficient soft tissue surrounding the knee
* Charcot's disease
* A fixed varus deformity (not passively correctable) of greater than 15 degrees
* A flexion deformity greater than 15 degrees
* Refuse to sign informed consent if it is required
* Patients that are not current residents of the United Kingdom

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 362 cases (121 investigational cases and 241 control cases) for primary efficacy and safety assessment (Primary Comparative Analysis Group); and exploratory assessment from one center in England.
  A total of approximately 1,000 investigational cases for "survivorship only" assessment from three centers.
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Composite Endpoint- Safety & Efficacy (Radiographic Success, American Knee Society Score, Absence of Revision / Removal / Unanticipated Adverse Device Affects) | 22+months
  Radiographic Success, American Knee Society Score, Absence of Revision / Removal / Unanticipated Adverse Device Affects

SECONDARY OUTCOMES:
Survivorship (Cementless Only) | 22+ Months
  Minimum 1,000 cases to assess survivorship of cementless components
American Knee Society Score | 0-16 Week, 6 Month, 12 Month
  Assessment of Function and Range of Motion; retrospective study- data will be collected if available
Oxford Knee Score | 0-16 Weeks, 6 Months, 12 Months, 22+ Months
  Retrospective study; data will be collected if available.
Adverse Events | Through 22+ Months Postop

CONTACTS AND LOCATIONS:
Overall Officials: Prof. David Murray, BA Hons, BChir, FRCS, MD, Principal Investigator — Nuffield Orthopaedic Centre; Prof. Hemant Pandit, MBBS, MS, DNB, FRCS, DPhil, Study Director — Nuffield Orthopaedic Centre

IPD SHARING:
Plan to Share IPD: Undecided
The primary analysis data is patient level data; collected in anticipation of potential PMA submission.